CLINICAL TRIAL: NCT00861354
Title: Home Monitoring for Atrial Fibrillation Using a Microlife Blood Pressure Monitor: Trial of Regular vs Irregualr Pulse for the Prevention of Stroke (TRIPPS 2.0)
Brief Title: Home Monitoring for Atrial Fibrillation Using a Microlife Blood Pressure Monitor
Acronym: TRIPPS
Status: Completed | Type: Observational
Sponsor: Microlife (Industry)
Responsible Party: Joseph Wiesel, MD, Microlife
Other Study IDs: tripps2
Record Dates: First submitted 2009-03-10; First posted 2009-03-13 (Estimated); Last update posted 2010-01-08 (Estimated); Status verified 2010-01

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; home blood pressure monitoring
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Microlife blood pressure monitor with AF detection (Microlife AFIB MLU3MQ1) — Monitoring heart rhythm daily for 30 days using the blood pressure monitor and the ECG recorder.
  Other Names: Microlife AFIB MLU3MQ1

SUMMARY:
This study assess the accuracy of a blood pressure monitor designed to detect atrial fibrillation. Subjects use the blood pressure monitor on a daily basis for 30 days and compare the readings to an ECG done at the same time.

ELIGIBILITY:
Inclusion Criteria: any of the following

* age 65 or older
* hypertension
* diabetes mellitus
* congestive heart failure
* previous stroke

Exclusion Criteria:

* permanent pacemaker
* impalantable defibrillator

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seen in a general medical practice.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the blood pressure monitor used for detecting atrial fibrillation compared to the electrocardiogram. | After final subject data is available.

SECONDARY OUTCOMES:
Assess subjects understanding of the use of the device for atrial fibrillation. | After final subject data is available.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Wiesel, MD, Principal Investigator
Locations (1):
- Joseph Wiesel, MD medical office, Flushing, New York, United States